CLINICAL TRIAL: NCT06458595
Title: A Phase I/II Study to Evaluate the Tolerability, Safety and Efficacy of KH658 Gene Therapy in Subjects With Neovascular Age-related Macular Degeneration (nAMD).
Brief Title: Safety and Tolerability of KH658 Gene Therapy in Subjects With Neovascular Age-related Macular Degeneration (nAMD)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chengdu Origen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KH658-40101
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-06

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KH658 (Experimental)
  Interventions: Drug: KH658

INTERVENTIONS:
Drug: KH658 — KH658 Ophthalmic Injection

SUMMARY:
KH658 is a adeno-associated virus (AAV) vector-based gene therapy for suprachoroidal space injection. The long-term, stable therapeutic protein after one time injection for nAMD could potentially reduce the treatment burden and maintain vision.

ELIGIBILITY:
Inclusion Criteria:

1. Are willing and able to sign the informed consent form (ICF);
2. Female and male aged 50 to 85 years (inclusive) with nAMD;
3. Have previously received anti-VEGF treatment for nAMD, with documented response to anti-VEGF therapy and a minimum of 2 anti-VEGF IVT injections in the study eye in the 6 months prior to screening;
4. Have a ETDRS BCVA letter score of 83 to 19 (approximately 20/25 to 20/400 Snellen equivalent) in the study eye at Screening;
5. Have a ETDRS BCVA letter score of ≥19 in the fellow eye at Screening;
6. Females must be at least 1 year postmenopausal.

Exclusion Criteria:

1. Have any other cause of CNV (such as pathological myopia, etc.) in the study eye; or non-nAMD disease in the study eye judged by the investigator that could impact macular examination or affect central vision (such as diabetic retinopathy, central retinal vein occlusion, etc.);
2. Any condition preventing visual acuity improvement in the study eye, e.g. fovea scar, fibrosis or atrophy;
3. Have a subretinal hemorrhage that is either 50% or more of the total lesion area, or blood is greater than 1.0 mm2 under the fovea in the study eye at screening;
4. Have any vitreous hemorrhage or history of vitreous hemorrhage in the study eye;
5. Presence of an implant (excluding intraocular lens), opacification of the refractive medium or miosis that affects fundus examination;
6. Have a history of or presence of retinal detachment or choroidal detachment in the study eye.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Tolerability and safety of KH658 in different dose levels | Week 4， Week 26
Change in BCVA letter | Week 26

SECONDARY OUTCOMES:
Incidence of adverse events and adverse reactions | Week 4， 26， 38， 54
Efficacy (BCVA, CRT) | Week 38， 54
Number of supplemental injections | Week 54
Annualized rate of supplemental injections | Week 54
Percentage of subjects free of rescue IVT therapy | Week 54

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China